CLINICAL TRIAL: NCT05210049
Title: Non-endoscopic Esophageal Sampling to Detect Barrett's Esophagus and Esophageal Cancer in Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1641950-1
Record Dates: First submitted 2021-12-16; First posted 2022-01-27 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Barrett Esophagus; GERD; Obesity; Esophageal Cancer
Keywords: Barrett Esophagus; Screening
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Obesity; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients undergoing routine screening via upper endoscopy (EGD) (Other): All enrolled patients will complete upper endoscopy for screening for Barrett's esophagus and esophageal adenocarcinoma.
  Interventions: Diagnostic Test: Esocheck/Esoguard

INTERVENTIONS:
Diagnostic Test: Esocheck/Esoguard — All enrolled patients will complete the Esocheck screening test. EsoCheck is a cell collection device that is designed to collect cells of a targeted region of the esophagus. The collected cell material is examined with a two marker panel combining methylated CCNA1 and VIM. These methylated markers have 95% sensitivity and 91% specificity for detecting BE and EAC with an AUC=0.95 in studies performed among white men. Diagnostic yield of this test among Veterans is unknown.

SUMMARY:
This study seeks to incorporate non-endoscopic detection method (Esocheck/Esoguard) in primary care practice and test whether this screening modality increases the positive predictive value of upper endoscopy and increases the detection of Barrett's esophagus and esophageal cancer.

DETAILED DESCRIPTION:
This study addresses prevention and early detection of esophageal adenocarcinoma (EAC). Prospectively collected Surveillance Epidemiology and End Results (SEER) data indicate that the incidence of esophageal adenocarcinoma (EAC) has increased more than 6-fold in the past four decades. The prognosis for patients with EAC is poor with less than 20% of patients surviving beyond 5 years. The veteran population is at increased risk for EAC and its precursor lesion, Barrett's esophagus (BE), due to increased prevalence of disease risk factors including advanced age, gastroesophageal reflux, caucasian race, male sex, smoking history, and obesity compared to the general population. Research has shown that veterans often present with an advanced cancer stage, despite opportunities to screen for BE in veterans with known risk factors. Therefore, there is an urgent clinical need to improve strategies for the detection and prevention of BE and EAC.

Currently, BE is diagnosed only when patients undergo endoscopy with esophagogastroduodenoscopy (EGD). However, due to the high cost of EGD and the lack of a randomized controlled trials supporting its efficacy, endoscopy to screen for BE is not routinely recommended. Current guidelines do recommend sedated EGD in patients with multiple BE risk factors, refractory GERD, or alarm symptoms. This strategy fails to detect BE in patients whose symptoms are well controlled with either over the counter medications or physician prescribed therapies. It also fails to detect BE in asymptomatic subjects who comprise 40% of those that develop EAC. Thus, less than 10% of esophageal adenocarcinomas are diagnosed as early stage lesions caught by surveillance of patients with previously detected BE. Ablative non-surgical therapies that have been developed for preventing cancer in patients with BE with high grade dysplasia over the past decade will have little impact and the 5 year survival for esophageal adenocarcinomas will remain a dismal 18% unless more effective programs for identifying BE and early EAC are developed.

The main hypothesis of this study is that incorporation of a non-endoscopic detection method in primary care practice will increase the positive predictive value of EGD and increase the detection of BE.

The objective of this study is to incorporate a novel unsedated BE screening method for veterans at risk for EAC into a primary care practice at a VA hospital.

Esocheck/Esoguard is a FDA approved device designed to sample the distal esophagus and analyze the collected material for presence of two methylated DNA markers.

The Specific Aims of this study are:

1. To determine sensitivity, specificity, positive and negative predictive value of Esocheck/Esoguard performed in routine practice for detecting BE in an at risk Veteran population
2. To compare the yield of detected BE using EGD alone vs. stepwise molecular diagnostics(Esocheck/Esoguard) and endoscopic screening strategy (EGD) in at risk Veteran population

ELIGIBILITY:
Inclusion Criteria:

Patients who have symptomatic GERD and also meet criteria for upper endoscopic screening for BE will be accrued. Eligible patients will include:

1. Adult Veterans > 40 and < 85 years old who have no prior EGD and can provide informed consent
2. No known coagulopathy, no known esophageal varices.
3. No significant dysphagia or odynophagia
4. Documented GERD or use of proton pump inhibitors (PPIs) for > 5 years
5. Meet ACG Clinical Guideline criteria for BE screening (that require presence of multiple risk factors 21). Eligible subjects to qualify must have will have GERD plus at least two additional risk factors for BE (white race, obesity defined as BMI > 30, male gender, smoking history, family history).

Exclusion Criteria:

1. Patients with known coagulopathy (INR > 1.5) will be excluded
2. Patients with known esophageal varices will be excluded.
3. Patients with significant dysphagia (unable to swallow solids) or odynophagia will be excluded

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Esocheck/Esoguard in a Veteran population | Through study completion, up to 2.5 years
  The accuracy of a test which reports the presence or absence of a condition, in comparison to a 'Gold Standard'

SECONDARY OUTCOMES:
Number/percentage of screened patients with diagnosis of Barrett's esophagus and/or esophageal adenocarcinoma | Through study completion, up to 2.5 years
  Compare diagnostic yield of EGD to diagnostic yield of Esocheck/Esoguard in Veterans
Cost of two screening strategies | Through study completion, up to 2.5 years
  Compare the cost of screening all enrolled patients by EGD alone vs. cost of selective screening by EGD in patients who have had a positive Esocheck/Esoguard test

CONTACTS AND LOCATIONS:
Overall Officials: Katarina B Greer, MD/MS, Principal Investigator — Louis Stokes Cleveland VA Medical Center
Locations (1):
- Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grady WM, Yu M, Markowitz SD, Chak A. Barrett's Esophagus and Esophageal Adenocarcinoma Biomarkers. Cancer Epidemiol Biomarkers Prev. 2020 Dec;29(12):2486-2494. doi: 10.1158/1055-9965.EPI-20-0223. Epub 2020 Oct 22. PMID 33093162
- [Background] Kaz AM, Wong CJ, Luo Y, Virgin JB, Washington MK, Willis JE, Leidner RS, Chak A, Grady WM. DNA methylation profiling in Barrett's esophagus and esophageal adenocarcinoma reveals unique methylation signatures and molecular subclasses. Epigenetics. 2011 Dec;6(12):1403-12. doi: 10.4161/epi.6.12.18199. PMID 22139570
- [Background] Moinova HR, LaFramboise T, Lutterbaugh JD, Chandar AK, Dumot J, Faulx A, Brock W, De la Cruz Cabrera O, Guda K, Barnholtz-Sloan JS, Iyer PG, Canto MI, Wang JS, Shaheen NJ, Thota PN, Willis JE, Chak A, Markowitz SD. Identifying DNA methylation biomarkers for non-endoscopic detection of Barrett's esophagus. Sci Transl Med. 2018 Jan 17;10(424):eaao5848. doi: 10.1126/scitranslmed.aao5848. PMID 29343623
- [Background] Tan WK, Sharma AN, Chak A, Fitzgerald RC. Progress in Screening for Barrett's Esophagus: Beyond Standard Upper Endoscopy. Gastrointest Endosc Clin N Am. 2021 Jan;31(1):43-58. doi: 10.1016/j.giec.2020.08.004. PMID 33213799
- [Derived] Greer KB, Blum AE, Faulx AL, Deming EM, Hricik LL, Siddiqui H, Wilson BM, Chak A. Nonendoscopic Screening for Barrett's Esophagus and Esophageal Adenocarcinoma in At-Risk Veterans. Am J Gastroenterol. 2025 Mar 1;120(3):545-553. doi: 10.14309/ajg.0000000000002962. Epub 2024 Jul 11. PMID 38989889